CLINICAL TRIAL: NCT00589394
Title: Analysis of the Mechanisms of Protective Humoral Immunity in Response to the Pneumococcal Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Miguel Park, Consultant, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 06-005905
Record Dates: First submitted 2007-12-28; First posted 2008-01-09 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Healthy
Keywords: pneumococcal vaccine; normal response; immunodeficiency; Healthy patients; Healthy Volunteers
MeSH Terms: conditions — Immunologic Deficiency Syndromes | interventions — Pneumococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- pneumococcal vaccination (Pneumovax) (Other): Intervention:
  Patients receive one dose of the Pneumovax vaccine. The 23 pneumococcal serotypes are measured before and after vaccination in order to measure response in a healthy population.
  Interventions: Biological: pneumococcal vaccination (Pneumovax)

INTERVENTIONS:
Biological: pneumococcal vaccination (Pneumovax) — pneumovax was given

SUMMARY:
The lack of clear guidelines and studies addressing the proper response to the pneumococcal vaccine (Pneumovax ®) has hampered our ability to diagnosis and care for our immunodeficiency patients. Should an age matched normal response range to the Pneumovax ® be established, it would have a profound impact in the diagnosis, safety and care of immunodeficiency patients. Moreover, characterizing the B cell compartments response to the Pneumovax ® may better delineate the mechanism of protective immunity from Pneumovax ® and provide an additional tool for the diagnosis and care for immunodeficiency patients.

DETAILED DESCRIPTION:
The ability to respond to a polysaccharide vaccine antigen is an integral part of evaluating a patient with immunodeficiency. The pneumococcal vaccine (Pneumovax ®) remains the only readily available and the most widely used unconjugated polysaccharide vaccine. Although the pneumococcal vaccine is widely used test the immune systems response to a polysaccharide antigen, no clear guidelines or studies exist to what is considered a proper response to the Pneumovax ®. Immunoglobulin M (IgM) memory B cells are thought to play an important role in protection against pneumococcal disease. It is not known to what extent the ability of B cells to be activated in response to pneumococcal vaccination contributes to protective immunity. To address these issues, the following two specific aims are proposed:

Specific Aim 1. Assess Immunoglobulin G (IgG) antibodies to pneumococcus pre- and post-pneumococcal immunization in healthy controls Specific Aim 2. Analysis of B cell subsets in blood of healthy controls pre-and post-pneumococcal immunization to identify changes in memory B cell, class switched and activated B cells.

ELIGIBILITY:
Inclusion Criteria:

* Patients from 20 to 70 years of age

Exclusion Criteria:

* Previous or current diagnosis of an immunodeficiency (primary and secondary)
* Previous or current diagnosis of a rheumatological disorders (Rheumatoid arthritis, Lupus, Sjögren, vasculitis), cancer, diabetes, active infection and/or other chronic diseases (multiple sclerosis, etc)
* Current or previous use (within that last 6 months) of systemic/inhaled corticosteroids, sulfasalazine, and other immunosuppressive agents (cyclosporin, methotrexate, CellCept) anti-convulsants (phenytoin, carbamazepine), gold, d-penicillamine, and anti-malarials (quinine, chloroquine, hydroxychloroquine)
* Pregnancy

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-07; Primary Completion 2008-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Assess IgG antibodies to pneumococcus pre- and post-pneumococcal immunization in healthy controls | 4-6 wks

SECONDARY OUTCOMES:
Analysis of B cell subsets in blood of healthy controls pre-and post-pneumococcal immunization to identify changes in memory B cell, class switched and activated B cells. | 4-6 wks

CONTACTS AND LOCATIONS:
Overall Officials: Miguel A. Park, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States